CLINICAL TRIAL: NCT06265441
Title: Comparison of IPACK Block with Adductor Canal Block Vs Adductor Canal Block Alone for Post Operative Analgesia Following Arthroscopic Knee Surgeries
Brief Title: Comparison of Pain Relief Post Knee Arthroscopy Using IPACK + Adductor Canal Block Vs. Adductor Canal Block Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS42/2024
Record Dates: First submitted 2024-02-07; First posted 2024-02-20 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A : Adductor canal block only (Experimental): Patients will receive Adductor canal block under ultrasound guide of 20 ml bupivacaine 0.25%
  Interventions: Procedure: Group A will receive adductor canal block after spinal anesthesia under a high-frequency ultrasound guidance in which the adductor canal is identified and 20 ml of 0.25% bupivacaine will be injected
- Group B : Adductor canal + IPACK block (Active Comparator): Patients will receive Adductor canal block and IPACK block under ultrasound guidance with 20 ml bupivacaine 0.25% for each block
  Interventions: Procedure: Group B will receive adductor canal block under ultrasound guide 20 ml bupivacaine 0.25% and IPACK block under direct visualization of ultrasound of 20 ml bupivacaine 0.25%

INTERVENTIONS:
Procedure: Group A will receive adductor canal block after spinal anesthesia under a high-frequency ultrasound guidance in which the adductor canal is identified and 20 ml of 0.25% bupivacaine will be injected — The patients in group A will receive adductor canal block after spinal anesthesia under a high-frequency ultrasound guidance (SonoSite™, Inc., Bothell, WA 98021, USA) in which the patients are placed in the supine position with the arms resting comfortably across the chest and the affected lower extremity is externally rotated. Adductor canal was identified beneath the sartorius muscle and 22-gauge 90-mm spinal needle is inserted from anterolateral to posteromedial direction at a point approximately at the junction between the middle and distal third of the thigh on the anteromedial femur, this location is called mid adductor canal, then 20 ml of 0.25% bupivacaine is injected in the canal
  Arms: Group A : Adductor canal block only
Procedure: Group B will receive adductor canal block under ultrasound guide 20 ml bupivacaine 0.25% and IPACK block under direct visualization of ultrasound of 20 ml bupivacaine 0.25% — The patients in Group B will receive adductor canal block as described in group A then IPACK block, in which the patients are placed in a supine position and knee is placed in position of 90° flexion. A low-frequency ultrasound probe is positioned in the popliteal crease 1 finger breadth above the patella, and a spinal needle is inserted from the medial aspect of the knee from anteromedial to posterolateral direction in a plane between the popliteal artery and the femur. The tip of the needle is placed 1-2 cm beyond the lateral edge of the artery, and 20 ml of 0.25% bupivacaine is injected while the needle is being withdrawn after negative aspiration.
  Arms: Group B : Adductor canal + IPACK block

SUMMARY:
In this study, the invistigators aim to compare postoperative analgesia effectiveness between combined interspace between the popliteal artery and posterior capsule of the knee block (IPACK) and Adductor canal block vs. Adductor canal block alone after Arthroscopic knee surgeries.

DETAILED DESCRIPTION:
Patients who fulfilled the inclusion criteria and agreed to participate in the study will be randomly divided into two groups using their computer-generated random numbers such that even numbers will be enrolled in group A for Adductor canal block alone and odd numbers will be enrolled in group B for Adductor canal block and IPACK block.

ELIGIBILITY:
Inclusion Criteria:

* Physical status: ASA 1 or 2
* Age group: 21-40 years.
* No sex predilection.
* Patients undergoing arthroscopic knee surgery under spinal anesthesia.

Exclusion Criteria:

* Patient refusal
* Physical status: ASA III or above.
* Patients with contraindications for spinal anesthesia.
* Patients with history of drug allergies to study drugs.
* Evidence of local infection at site of injection.
* Neuromuscular pathology (example: - Multiple Sclerosis)

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Assessment of pain using the visual analogue scale (VAS) at 2 hours, 4 hours, 6 hours, and 8 hours after the completion of the surgical procedure and skin closure. | 8 hours
  Visual analogue scale (VAS) (scale 0-10, where 0 = no pain and 10 = worst imaginable pain). All the patients will have the VAS score explained and taught for self-assessment of pain at the time of enrolment for the study.

SECONDARY OUTCOMES:
Total pethidine consumption | 24 hours
  Total pethidine consumption (in mg.) over 24-hour period post-operative
The time till first analgesic requirement | as requested by patient
  The time (in hours) after finishing of ultrasound guided IPACK or Adductor canal blocks till the patient's requirement for first analgesia postoperative in ward. (All patients will receive intravenous pethidine (30mg) when VAS > 4 at any time of assessment)
The number of steps | 24 hours
  ambulation distance assessed by the number of steps walked by the patient 24 hours after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Morsi, M.B.B.CH, Principal Investigator — Anesthesia resident, Ain shams university
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt